CLINICAL TRIAL: NCT00003252
Title: A Phase IV Open Label Study of the Effects of a Five Minute Infusion Time for Ethyol (Amifostine) in Patients Undergoing Chemotherapy
Brief Title: Amifostine in Treating Patients With Cancer Who Have Neurological Changes Caused by Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush North Shore Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000066134; RNSMC-AM9702; ALZA-RNSMC-AM9702; NCI-V98-1390
Record Dates: First submitted 1999-11-01; First posted 2004-09-10 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2000-04

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Amifostine

INTERVENTIONS:
Drug: amifostine trihydrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase IV trial to study the effectiveness of amifostine in treating patients with cancer who have neurological changes caused by chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and tolerability of administering amifostine by intravenous infusion over 5 minutes in cancer patients undergoing chemotherapy.

OUTLINE: This is an open label, controlled study. Patients receive intravenous amifostine over 5 minutes 30 minutes prior to chemotherapy. Patients are followed for one month post treatment.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven cancer No brain or other CNS metastases (including prior treated metastases)

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-1 Life Expectancy: Not specified Hematopoietic: Not specified Hepatic: No grade 3 or greater hepatic dysfunction Renal: No hypercalcemia Cardiovascular: No uncontrolled hypotension Other: Not pregnant or nursing Effective contraceptive method must be used by fertile patients No psychosis No severe concurrent illness other than neoplasia No epileptic seizures during the previous year, migraines, gastrointestinal obstructions, or other causes of vomiting No prior or concurrent amifostine contraindications No prior known contraindications or sensitivity to dexamethasone, granisetron, ondansetron, prochlorperazine, diphenhydramine, cimetidine, or magnesium

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No prior estrogen within 24 hours of amifostine therapy Radiotherapy: Not specified Surgery: Not specified Other: No prior alcohol, disulphiram, tetracycline, or erythromycin within 24 hours of amifostine therapy No prior antiemetics such as benzodiazepines, antipsychotics, anticonvulsants, or antihistamines within 24 hours of amifostine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-12; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward H. Kaplan, MD, Study Chair — Rush North Shore Medical Center
Locations (1):
- Rush North Shore Medical Center, Skokie, Illinois, United States